CLINICAL TRIAL: NCT04821323
Title: A Phase 0 Platform Study Exploring the Use of Challenge Agents in Healthy Volunteers
Brief Title: A Study Exploring the Use of Challenge Agents in Healthy Volunteers - Intervention Specific Appendix
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CR108965; NOPRODPCNAP0001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-03-17; First posted 2021-03-29 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Healthy
MeSH Terms: interventions — Indomethacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Indomethacin Challenge (Experimental): Participants will receive challenge agent as two single oral doses of Indomethacin, one on Day -1 and one on Day 1. In addition, participants will receive lactulose-mannitol solution on Day -4 (baseline) and on Day 1 (post Indomethacin challenge).
  Interventions: Drug: Indomethacin; Diagnostic Test: Lactulose-mannitol

INTERVENTIONS:
Drug: Indomethacin — Indomethacin capsules will be administered orally.
Diagnostic Test: Lactulose-mannitol — Lactulose-mannitol solution will be administered orally.

SUMMARY:
The purpose of this study is to characterize the disruption of intestinal barrier as a result of indomethacin challenge in healthy volunteers using an orally administered lactulose-mannitol test.

ELIGIBILITY:
Inclusion Criteria:

* healthy on the basis of physical examination, medical history, and vital signs, and 12-lead electrocardiogram (ECG) performed at screening. Any abnormalities, must be consistent with the underlying illness in the study population and this determination must be recorded in the participant's source documents and initialed by the investigator
* healthy on the basis of clinical laboratory tests performed at screening. If the results of the serum chemistry panel, hematology, or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator
* must be a non-smoker (not smoked for at least 6 months prior to screening) and has not used nicotine-containing products (example, nicotine patch) for 3 months prior to screening
* A woman must be: a) not of childbearing potential; b) Of childbearing potential and practicing a highly effective method of contraception (failure rate of less than (<1) percent (%) per year when used consistently and correctly) and agrees to remain on a highly effective method while receiving study intervention and until the end of the intervention cohort. The investigator should evaluate the potential for contraceptive method failure (example, noncompliance, recently initiated) in relationship to the first dose of study intervention
* A woman of childbearing potential must have a negative highly sensitive serum (beta-human chorionic gonadotropin [beta-hCG]) at screening and a negative urine pregnancy test prior to study intervention administration on Day -4

Exclusion Criteria:

* history of liver or renal insufficiency; significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances
* history of any type of immunodeficiency or autoimmune disease or disease treatment associated with immune suppression or lymphopenia. These include but are not limited to bone marrow or organ transplantation, lymphoproliferative disorders, T- or B-cell deficiency syndromes, splenectomy, functional asplenia and chronic granulomatous disease
* has an active, acute or chronic infection
* has a history of inflammatory bowel disease (IBD), celiac disease, or gastrointestinal diseases (GI) surgery, excluding appendectomy and cholecystectomy
* has known allergies, hypersensitivity, or intolerance to aspirin or nonsteroidal anti-inflammatory drugs (NSAIDs)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2021-05-07 (Actual)

PRIMARY OUTCOMES:
Longitudinal Change From Baseline in Lactulose/Mannitol Ratio in the Urine Following Indomethacin Challenge | Baseline, Up to 14 days
  Longitudinal change from baseline in L/M ratio in the urine following indomethacin challenge will be assessed. L/M ratio in urine is a useful and noninvasive marker for the evaluation of intestinal permeability in the urinary excretion of these nonmetabolized sugars.
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) | Up to 6 weeks
  An adverse event (AE) is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. TEAEs are defined as AEs with onset or worsening on or after date of first dose of study treatment.
Number of Participants with Treatment-Emergent Serious Adverse Events (TE-SAEs) | Up to 6 weeks
  TE-SAEs is defined as any untoward medical occurrence with a reasonable possibility that it is caused by the study intervention that: Is life-threatening (example; leads to stroke or non-fatal pulmonary embolism); Requires inpatient hospitalization or prolongation of existing hospitalization; Results in persistent or significant disability/incapacity; Results in other clinically significant sign(s) or symptom(s), (example; clinically asymptomatic brain microhemorrhages); or Results in death.

SECONDARY OUTCOMES:
Longitudinal Change From Baseline in Selected Biomarkers Following Indomethacin Challenge | Baseline, Up to 14 days
  Change from baseline in selected biomarkers levels (example: Lactulose-mannitol, C-reactive protein [CRP], calprotectin, Et cetera [etc.]) using analysis methods such as liquid chromatography/mass spectrometry, immunoturbidimetry, enzyme-linked immunosorbent assay (ELISA), etc., as a result of the indomethacin challenge.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Clinical Pharmacology Unit, Merksem, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency